CLINICAL TRIAL: NCT06872632
Title: EFFETTI DELLA COMPLESSITÀ E MULTIMORBIDITÀ SUGLI ESITI CLINICI NEL PAZIENTE INTERNISTICO OSPEDALIZZATO: STUDIO MULTICENTRICO, OSSERVAZIONALE E PROSPETTICO - EFFECTS of COMPLEXITY and MULTIMORBIDITY on CLINICAL OUTCOMES in HOSPITALIZED INTERNAL MEDICINE PATIENTS: a MULTICENTER, OBSERVATIONAL and PROSPECTIVE STUDY
Brief Title: How Complexity and Multiple Illnesses Affect Hospitalized Patients' Health: a Multicenter Study
Status: Recruiting | Type: Observational
Sponsor: Società Italiana di Medicina Interna (Other)
Responsible Party: Sponsor
Other Study IDs: 207/2023/OSS/AOUMO
Record Dates: First submitted 2025-02-25; First posted 2025-03-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Complexity and Multiple Illnesses of Adult Hospitalized Internal Medicine Patient

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this observational study is to evaluate the association between complexity and multiple illnesses of adult hospitalized internal medicine patient and mortality. The observational study will also evaluate the association between pre-existing factors at hospitalization and clinical outcomes such as mortality, length of hospital stay, intensity of care (transfer to units with higher clinical intensity), complications and rehospitalization.

For data collection, four index weeks will be identified during the year in which the participating Centers will have to sequentially enroll all the participants who will be admitted to the Internal Medicine units, until reaching, for each index week, 10 participants for each of the Participating Centers.

Each enrolled participant will undergo a 12-month follow-up. The study foresees the enrollment of 2326 participants.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of legal age (age >= 18 years).
2. Informed consent according to Italian law.

Exclusion Criteria:

* No specific exclusion criteria were identified.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult hospitalized internal medicine patient
Sampling Method: Non-Probability Sample
Enrollment: 2326 (Estimated)
Dates: Start 2024-06-24 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
to evaluate the correlation between clinical complexity/multimorbidity of the hospitalized internal medicine patient, defined by the Cumulative Illness Rating Scale (CIRS), and mortality. | 12 months
  to evaluate the correlation between clinical complexity/multimorbidity of the hospitalized internal medicine patient, defined by the Cumulative Illness Rating Scale (CIRS), and mortality. Cumulative Illness Rating Scale: severity index (minimum value is 1, maximum value is 5), comorbidity index (minimum value is 0, maximum value is 13). Higher scores mean worse outcome.

SECONDARY OUTCOMES:
to evaluate the correlation between pre-existing factors at hospitalization and clinical outcomes - to evaluate the association between disease severity parameters and clinical outcomes | 12 months
  * to evaluate the correlation between pre-existing factors at hospitalization, such as polypharmacy, age, prevalent chronic diseases (e.g. heart failure, respiratory failure and pneumonia, decompensated diabetes, etc.) and clinical outcomes such as mortality, length of hospital stay, intensity of care (transfer to units with higher clinical intensity), complications and rehospitalization
  * to evaluate the association between disease severity parameters (e.g. biohumoral, score, etc.) and clinical outcomes.

CONTACTS AND LOCATIONS:
Locations (12):
- Italy (12):
  - AOU Policlinico di Bari- Unità Operativa di Medicina Interna "Guido Baccelli, Bari, Italy
  - Azienda Ospedaliero Universitaria di Bologna Policlinico S. Orsola - Malpighi- UO Medicina interna, malattie epatobiliari e immunoallergologiche, Bologna, Italy
  - ASST degli Spedali Civili di Brescia- Medicina Generale 2, Brescia, Italy
  - Azienda Ospedaliero-Universitaria S. Anna di Ferrara- Clinica Medica, Ferrara, Italy
  - Ospedale Santa Maria Annunziata, Bagno a Ripoli, Firenze- Medicina 1, Florence, Italy
  - AOU G. Martino- UOC Medicina Interna, Messina, Italy
  - ASST Fatebenefratelli Sacco, Ospedale Luigi Sacco- Struttura Complessa di Medicina Interna, Milan, Italy
  - AOU Modena - Policlinico di Modena - S.C. Medicina Interna, Modena, Italy
  - Azienda Ospedaliera Universitaria Federico II, Napoli- UOC Medicina Interna ad indirizzo metabolico e riabilitativo, Napoli, Italy
  - Ospedale Maggiore della Carità di Novara- SCDU Medicina Interna 1, AOU Maggiore della Carità, Novara, Italy
  - Policlinico Universitario Campus Bio-Medico di Roma- UOC Medicina Interna, Roma, Italy
  - Azienda Ospedaliero-Universitaria Sant'Andrea- UOC Medicina Interna, Roma, Italy